CLINICAL TRIAL: NCT04501328
Title: A Randomized Controlled Trial of Coaching Into Care With VA-CRAFT to Promote Veteran Engagement in PTSD Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency); Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 19-031
Record Dates: First submitted 2020-08-03; First posted 2020-08-06 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Stress Disorders, Post-traumatic
Keywords: Stress Disorders, Post-traumatic; Internet-Based Intervention; Telemedicine; Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Coaching Into Care plus VA-CRAFT consists of four 45-min. telephone coaching calls over 8-12 weeks, delivered by a coach following a manual. Calls focus on supporting and holding the participant accountable for using the VA-CRAFT for PTSD web-based course. This course is based on Community Reinforcement and Family Training (CRAFT) which is intended to help family members of Veterans with PTSD who are resistant to seek treatment for PTSD to initiate care as well as promote the family member's wellbeing and improve their relationship with the Veteran. Calls are designed to: 1) help participants maintain motivation to complete VA-CRAFT lessons in a timely fashion by using reinforcement and motivational techniques; 2) consolidate information and implement skills that they are learning in the course through lesson review, role plays, and problem solving; and, 3) normalize and validate the challenges of having a loved one with PTSD who is reluctant to seek care (i.e., supportive caring).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CIC+VA-CRAFT (Experimental): Coaching Into Care plus VA-CRAFT consists of four 45-min. telephone coaching calls over 8-12 weeks, delivered by a coach following a manual, while participants are completing the VA-CRAFT for PTSD web-based course.
  Interventions: Behavioral: CIC+VA-CRAFT
- CIC (Active Comparator): Coaching Into Care is an existing national VA program that provides telephone consultation and coaching to family members of Veterans with mental health needs who want to help connect them with mental health care by providing referrals, educational information, and a unique coaching service to help callers talk to their Veterans about their decision to seek care.
  Interventions: Behavioral: CIC

INTERVENTIONS:
Behavioral: CIC+VA-CRAFT — CIC+VA-CRAFT consists of four 45-min. telephone coaching calls over 8-12 weeks, delivered by a coach following a manual, while participants are completing the VA-CRAFT for PTSD web-based course.
  Other Names: Coaching Into Care plus VA-CRAFT
  Arms: CIC+VA-CRAFT
Behavioral: CIC — Coaching Into Care is an existing national VA program that provides telephone consultation and coaching to family members of Veterans with mental health needs who want to help connect them with mental health care by providing referrals, educational information, and a unique coaching service to help callers talk to their Veterans about their decision to seek care.
  Other Names: Coaching Into Care
  Arms: CIC

SUMMARY:
Posttraumatic stress disorder (PTSD) afflicts many war Veterans, but often they are reluctant to seek help despite availability of effective treatments. Family members are key sources of support who can help encourage such Veterans to initiate mental health services. Toward that goal, VA provides telephone coaching to family members through its Coaching Into Care (CIC) program to help get their Veterans into care. While CIC enjoys high caller satisfaction, it has shown only modest success getting Veterans into care. Blended interventions that include professional support and technology-based interventions offer promise for improving effectiveness of services. Therefore, this study tests an intervention that blends CIC calls with a web program called VA Community Reinforcement and Family Training (VA-CRAFT). VA-CRAFT is a translation of an empirically-validated model intended to help Veterans by training their family members to effectively promote care-seeking. If successful, this approach will support families and help more Veterans receive needed mental health care for PTSD.

DETAILED DESCRIPTION:
Posttraumatic Stress Disorder (PTSD) is a highly prevalent, potentially debilitating condition afflicting many war Veterans. While efficacious treatments are available, most individuals with PTSD do not receive any mental health care. VA faces an ongoing challenge of engaging Veterans with PTSD in effective services. Recognizing the powerful influence of families on Veteran wellbeing, VA has called for increased involvement of family members in the care of Veterans with PTSD. In response, VA has created a national telephone-based support service called Coaching Into Care (CIC) to work with family members of Veterans with mental health problems who are reluctant to seek treatment. Program evaluation data show that CIC is highly valued by callers, but that only about 25% of callers with Veterans not already in care, report that their Veteran sought care over the next six months. The proposed study is a test of an innovative approach to improve outcomes by blending coaching calls with a web-based program called VA Community Reinforcement and Family Training (VA-CRAFT). VA-CRAFT is a translation of an empirically-validated model intended to help Veterans by training and supporting their family members to better care for themselves, more effectively manage their relationships, and have effective care-seeking conversations with their Veterans.

Preliminary work suggests that VA-CRAFT may be a powerful adjunct for CIC services. In a prior HSR&D-funded pilot, the investigators' team found that family members who completed the relatively brief VA-CRAFT course alone (without any coaching) had greater decreases in caregiver burden than wait-list controls. However, qualitative interviews also suggested that participants often did not raise the issue of treatment with their Veteran loved one due to not believing such a conversation would be successful. The investigators developed CIC+VA-CRAFT with the goal of capitalizing on the strengths of both approaches (CIC and VA-CRAFT) and increasing family members' motivation, perceived ability to have treatment-seeking conversations with the Veteran, and success at engaging their Veterans in care. Initial findings from a second, NC-PTSD-funded pilot suggest that this brief, blended intervention is feasible, acceptable, and potentially more effective than CIC alone in enhancing Veteran mental health treatment initiation.

Primary Objective: The primary objective is to investigate the effectiveness of CIC+VA-CRAFT in improving Veteran treatment initiation above CIC only, without compromising the high caller satisfaction of the CIC program. To accomplish this, the investigators will use a two-group randomized controlled trial. Spouse/partners who believe their Veteran needs PTSD treatment will be randomized to CIC+VA-CRAFT or CIC only (i.e., TAU). Assessments will occur at baseline, post-treatment (month 3), and follow-up (month 6). To maximize generalizability of findings to the intended population, recruitment will use targeted social media advertising and referrals from the existing CIC program. Specific aims are:

Aim 1: Determine the effectiveness of CIC+VA-CRAFT for Veteran mental health service initiation. The investigators hypothesize that spouse/partners in CIC+VA-CRAFT will report higher rates of mental health service initiation for their Veterans than will participants in the CIC only condition.

Aim 2: Investigate caller satisfaction with CIC+VA-CRAFT relative to CIC only. The investigators hypothesize that satisfaction with CIC+VA-CRAFT will be non-inferior to satisfaction with the CIC program.

Aim 3: Conduct a process evaluation to inform potential future implementation of CIC+VA-CRAFT. Qualitative interviews with spouse/partners, their Veterans, and study and CIC coaches, will be used to inform future implementation of the CIC+VA-CRAFT intervention into the CIC program.

Exploratory Aims:

1. Explore potential within-condition improvements and between-condition changes on spouse/partner and family outcomes. The investigators will test for these effects on measures of caregiver burden, psychological distress, quality of life, and family conflict and cohesion.
2. Explore potential intervention mediators and moderators of Veteran mental health treatment initiation. The investigators will explore if self-efficacy, outcome expectancy, and treatment conversations mediate the effect of the intervention on mental health treatment initiation. Demographic variables, perceived Veteran symptomatology, and partner symptomatology will be explored as moderators of the effect of the intervention.

The long-term goal of this research is to establish an efficacious, efficient, scalable, and satisfying family outreach intervention that will significantly increase mental health service initiation among a high priority Veteran population while addressing the needs of their primary supporters, their family members. This proposal has been developed in collaboration with the existing VA CIC and VA-CRAFT programs and involves the leadership of these programs to facilitate the blended intervention's rapid dissemination should the trial prove successful.

ELIGIBILITY:
Inclusion Criteria:

The target population consists of partners and first-degree family members who are in regular contact with a Veteran from any service era who believe that their Veteran is suffering from significant symptoms of PTSD and in need of mental health care.

Inclusion criteria are:

* reporting being in an intimate relationship (dating, engaged, or married) with a Veteran or a first degree family member of a Veteran
* reporting that their Veteran is not engaged in mental health care and has not been for the past 6 months
* reporting perceived symptoms of PTSD in their Veteran
* reporting frequent contact with their Veteran (some verbal or face-to-face contact for 36 of the past 90 days)
* having regular access to the Internet and a telephone; and 6) being 18 years of age or older

Exclusion Criteria:

* reporting by the potential participant that they are subject to domestic violence and may not feel safe engaging in CIC+VA-CRAFT activities
* we will exclude partners reporting severe intimate partner violence on the brief Conflict Tactics Scale 2 Short Form with their Veteran in the past 6 months

  * appropriate referrals for those excluded based on recent intimate partner violence will be provided

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Veteran Mental Health Service Utilization Change | 3 and 6 months post-randomization
  Veteran mental health service initiation as reported by the enrolled partner. This will be operationalized dichotomously (whether any mental health services are initiated) for VA and non-VA services for the 3- and 6-month periods following randomization.
Client Satisfaction Questionnaire (CSQ; Attkisson et al., 1979) | 3 months post-randomization
  This 8-item measure assesses general client satisfaction at post-treatment stage for the intervention delivered in the study. The Client Satisfaction Questionnaire is a self-report measure with each item score ranging from 1 to 4. The total score is derived from summing all items ranging from 1 to 32, with higher scores reflecting greater program satisfaction.

SECONDARY OUTCOMES:
Montgomery Borgatta Caregiver Burden Scale( Montgomery & Borgatta, 1985) | 3 and 6 months post-randomization
  This 22-item measure assesses the change in the objective burden, subjective stress burden, and subjective demand burden of caregiving over twelve weeks. Final score is the total sum of each item, where each item score ranges from 0 to 4 with the final score ranging from 0 to 88. The total raw score will indicate either little or no caregiver burden (0 to 20), mild to moderate caregiver burden (21 to 40), moderate to severe caregiver burden (41 to 60) or severe caregiver burden (61-88).
World Health Organization - Quality of Life (Brief; WHOQOL; World Health Organization, 1996)) | 3 and 6 months post-randomization
  This 26-item self-report measure assesses the change in four domains of quality of life over twelve weeks: physical health, psychological health, social relationships, and environment. Each item score ranges between 1 to 5. To assess each domain, total scores for items measuring that domain are further calculated and transformed into a 0 to 100 scale. Domain scores are in positive direction, where higher scores indicate higher quality of life.
Brief Symptom Inventory (BSI; Derogatis, 2000) | 3 and 6 months post-randomization
  This 18-item self-report measure assesses the change in psychological distress and psychiatric symptoms over twelve weeks. Each item score ranges between 0 to 5, where final score of all items are aggregated and transformed into a t-score for three subscales on the Global Severity Index (GSI): somatization, depression and anxiety. Higher t-score for each subscale on the GSI indicates clinically significant symptoms.
Family Environment Scale (FES; Moos, 1974) | 3 and 6 months post-randomization
  The 20-item self-report measure assesses the change in general familial relationship functioning, with subscales measuring Cohesion and Conflict over twelve weeks. Each item is a 'Yes' or 'No' item with a scoring or 1 and 0, respectively. Subscales are scored by summing scores for items measuring their component subscale, resulting in two subscale scores. The subscale scores are then used to categorize families' social climate.

CONTACTS AND LOCATIONS:
Overall Officials: Eric R Kuhn, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA; Steven L. Sayers, PhD, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuhn E, Sayers S, Zimmerman L, Mackintosh MA, Owen JE, Rosen CS, Meis LA, Hagedorn HJ, Erbes CR. Promoting mental health treatment initiation of veterans with PTSD using internet-based family training and telephone coaching: Protocol for a randomized controlled trial. Contemp Clin Trials. 2025 Jul;154:107929. doi: 10.1016/j.cct.2025.107929. Epub 2025 May 2. PMID 40320070

DOCUMENTS (1):
  • Informed Consent Form (2025-02-28): https://cdn.clinicaltrials.gov/large-docs/28/NCT04501328/ICF_000.pdf